CLINICAL TRIAL: NCT07047989
Title: Safety, Tolerability and Immunogenicity Study of NWRD09 in HPV16 Related Cervical High-grade Squamous Intraepithelial Lesions (HSlL)
Brief Title: NWRD09 for HPV-16 Related Cervical HSIL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Newish Biotech (Wuxi) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NWRD09-102
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: High-grade Squamous Intraepithelial Lesion (HSIL)
Keywords: NWRD09; mRNA vaccine; HPV16; HSIL
MeSH Terms: conditions — Squamous Intraepithelial Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose1-3 of NWRD09 (Experimental): Patients will be assigned to three dose groups. Each patient will be administered NWRD09 by intramuscular injection. The Maximum Tolerated Dose of NWRD09 will be determined by the classical 3+3 dose escalation schedule. The number of patients will be ranged from 9 to 18.
  Interventions: Biological: NWRD09 injection

INTERVENTIONS:
Biological: NWRD09 injection — NWRD09 administered by intramuscular injection

SUMMARY:
This is a single-arm, open label, multi-center clinical study to evaluate the safety, tolerability and immunogenicity HPV16 targeted mRNA therapeutic vaccine (NWRD09) in HPV16 related cervical high-grade squamous intraepithelial lesions (HSlL).

DETAILED DESCRIPTION:
This study is divided into three dose groups. Each patient will be administered NWRD09 by intramuscular injection at week 0,2,4 and12. The Maximum Tolerated Dose of NWRD09 will be determined by the classical 3+3 dose escalation schedule. The number of patients will be ranged from 9 to 18.

The subjects shall continue to receive safety follow-up until 28 days after the third administration. Colposcopy and biopsy were performed at week 24.

This study will select 1-2 dose levels for subject expansion based on the dose escalation phase, to further evaluate the safety, tolerability, immunogenicity, and efficacy of NWRD09 in HPV16 related cervical HSIL patients.

ELIGIBILITY:
Inclusion Criteria:

Patients had to meet all of the following inclusion criteria:

1. Women aged between 18 and 65 years.
2. HPV16-positive patients with histologically confirmed cervical HSlL.
3. Colposcopic examination should be adequate, enabling clear visualization of the entire squamocolumnar junction(SCJ), as well as the full extent of acetowhite staining or suspected cervical intraepithelial neoplasia (ClN) lesions, including the upper boundary of the lesion.
4. Major organ functions were normal within 1 week before the first NWRD09 administration: 1) Blood routine: Hemoglobin (Hb) ≥100 g/L; Platelet count (PLT) ≥75×109/L; 2) The liver: Total bilirubin (TB) ≤1.5× upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; Plasma albumin ≥30 g/L; 3)Kidney: Serum creatinine (Scr) ≤1.5×ULN, or creatinine clearance ≥40mL/min (Cockcroft-Gault);
5. For premenopausal women of child bearing potential, a blood pregnancy test must yield a negative result within 7 days prior to the first administration of the investigational drug; eligible subjects with reproductive capacity, as well as their spouses/partners, must agree to use effective contraceptive measures during the trial period or for at least 6 month safter the end-of-study visit (Week 24).
6. Have fully understood the study and voluntarily signed the ICF, have good communication with the investigator, and are able to complete all treatments, examinations, and visits stipulated in the study protocol.

Exclusion Criteria:

Patients with any of the following were excluded from the study:

1. Any histologically confirmed adenocarcinoma or adenocarcinoma in situ (AIS) or invasive cancer.
2. Pregnant, breastfeeding, or planning to conceive during the study period.
3. Participated in another clinical trial or is in the observation period of another clinical trial within 30 days prior to screening.
4. Continuous (more than 1 week) use of corticosteroids (equivalent to >10 mg/day of prednisone) within 30 days prior to screening, except for hormone replacement therapy and local administration such as inhaled or ocular treatments.
5. Continuous (more than 1 week) use of immunosuppressants (e.g., cyclosporine, tacrolimus, azathioprine, 6-mercaptopurine, and anti-lymphocyte globulin) within 30 days prior to screening.
6. Received any non-live/live vaccine injection within 4 weeks prior to the first dose of NWRD09.
7. Any history of therapeutic HPV vaccination (previously approved preventive HPV vaccination is acceptable).
8. Received treatment HSIL within 4 weeks prior to the first dose of NWRD09.
9. Prohibited: Use of blood/blood-derived products (e.g., immunoglobulins) within 3 months before first dose or intended use during the study.
10. History of immunodeficiency or autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis).
11. Current or anticipated use of disease-modifying antirheumatic drugs (e.g., azathioprine, cyclophosphamide, cyclosporine, methotrexate) and biological agents (e.g., infliximab, adalimumab, etanercept) during the study.
12. History of solid organ or bone marrow transplantation.
13. Past or current malignancies, except for adequately treated and completely cured ductal carcinoma in situ of the breast, basal cell carcinoma of the skin, superficial bladder tumors, or any other malignancies cured more than 5 years before entering the study.
14. Uncontrolled severe infections (>Grade 2 NCI-CTCAE adverse events, version 5.0).
15. Patients who test positive for any of the following: hepatitis C virus (HCV)antibody, human immunodeficiency virus (HlV) antibody, or syphilis treponema antibody; except those with abnormal hepatitis B serology (i.e., positive for hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb]) but meet one of the following criteria:

1)HBV-DNA ≤2,500 copies/mL or ≤ 500lU/mL, or 2)HBV-DNA within the normal reference range of the testing center. 16.History of severe or multiple hypersensitivity to drugs or pharmaceutical preparations.

17.Severe dysfunction of other organs or heart and lung diseases. 18.History of definite neurological or psychiatric disorders, including epilepsy or dementia.

19.History of drug abuse or alcoholism. 20.Patients deemed unsuitable to participate in this clinical trial by the investigator.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety | To week 24
  All adverse events (AE) will be determined based on the rate and severity grade of events, including incidence and severity of serious adverse events (SAE) (according to NCI-CTCAE Standard version 5.0 of common Terms for Adverse Events).
Dose-limiting toxicity (DLT) | Within 28 days of the third dosing
  It would be determined based on the rate and severity grade of events or abnormalities through evaluating systemic or local adverse events, clinical laboratory test results, vital signs that is definitely, probably, or possibly related to the test drug occurring within 28 days of the third dosing will be classified as DLT during dosing climb.

SECONDARY OUTCOMES:
Immunogenicity | Week 4、8、16、24、48
  Immunologic reactogenicity by measuring HPV16 specific T cell response (IFN-γ ELISPOT) and anti HPV16 antibodies (ELISA) in blood samples
Histopathology outcome and HPV Viral clearance | Week 24.
  Number of subjects with virologically-proven clearance of HPV 16 and number of subjects with histopathological regression of cervical lesions to CIN 1 or normal
The recommended phase II dose (RP2D) | Week 24
  The recommended phase II dose (RP2D) was selected on the basis of tolerability during the safety expansion.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided